CLINICAL TRIAL: NCT02958631
Title: Comparison of Blood Pressure Lowering Effect Between Fimasartan and Losartan in the Hypertensive Patient During Night and Early Morning Time
Brief Title: Comparison of Blood Pressure Lowering Effect Between Fimasartan and Losartan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Sang Min Park, MD, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEFILONE Study
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fimasartan (Experimental): Fimasartan 60mg, QD
  Interventions: Drug: Fimasartan
- Losartan (Active Comparator): Losartan 50mg, QD
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Fimasartan
  Other Names: Kanarb
  Arms: Fimasartan
Drug: Losartan
  Other Names: Cozaar
  Arms: Losartan

SUMMARY:
Comparison of blood pressure lowering effect between Fimasartan and Losartan in the hypertensive patient during night and early morning time

ELIGIBILITY:
Inclusion Criteria:

* Subject don't have Anti-hypertensive drug or who stop Anti-hypertensive drug during 2 weeks
* Office BP: over siSBP 140mmHg or si DBP 90mmHg
* 24hr ABPM: SBP 130mmHg or DBP 80mmHg (24 hour Average)

Exclusion Criteria:

* Pregnant, trying to become pregnant or breast feeding
* Subject has Secondary Hypertension
* White coat Blood Pressure (Normal result of 24 hour ABPM)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Lowering Effect through 24 ABPM | 24 hour
  comparing blood pressure lowering effect between night and early morning

IPD SHARING:
Plan to Share IPD: No